CLINICAL TRIAL: NCT03995342
Title: The Correlation and Intervention of Intestinal Flora and Frailty in the Elderly
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaoming-1, Director of geriatrics, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY20192015-F-1
Record Dates: First submitted 2019-06-10; First posted 2019-06-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Frailty Syndrome
Keywords: frailty, flora
MeSH Terms: conditions — Frailty | interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exprimental: Inulin (Experimental): Inulin 15 grams after dissolution by mouth， every morning for three months.
  Interventions: Dietary Supplement: Inulin
- Active comparator: maltodextrin (Placebo Comparator): Placebo (maltodextrin) 15grams after dissolution by mouth， every morning for three months.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin 15 grams after dissolution by mouth， every morning for three months.
  Arms: exprimental: Inulin
Dietary Supplement: Maltodextrin — Placebo (maltodextrin) 15g/d，Oral administration after dissolution15g/d，Oral administration after dissolution
  Other Names: Placebo
  Arms: Active comparator: maltodextrin

SUMMARY:
The study aim to evaluate the improvement and correlation of soluble dietary fiber (prebiotics) in the frailty of elderly people by a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
100 healthy controls, 100 pre-frailty and 100 frailty elderly will be included. the healthy controls will be received no intervention. The pre-frailty will be randomized at a 1：1 ratio to receive prebiotics (inulin) or placebo (maltodextrin) . The degree of improvements and correlation in frailty will be evaluated three months later.Similarly,the frailty also will be randomized at a 1：1 ratio to receive prebiotics (inulin) or placebo (maltodextrin). The degree of improvements and correlation in frailty will be evaluated three months later.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years;
* Can get up from a chair and walk 6 meters
* Clearly consciousness, able to read or use words to express and communicate without difficulty
* Agree and accept the study plan

Exclusion Criteria:

* Acute and chronic inflammatory disease of the intestine within 3 months
* Use of antibiotics, probiotics, prebiotics or synthetics, laxatives or diarrhea medications, proton pump inhibitors or gastric motility drugs within 1 month
* Dementia
* mental illness or blindness
* acute infection
* cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of frailty | 3 months
  Frailty will be diagnosed according to Fried criteria

SECONDARY OUTCOMES:
Diversity analysis of intestinal flora | 3 months
  Change of diversity analysis of intestinal flora

CONTACTS AND LOCATIONS:
Overall Officials: Wang xiao ming, Study Chair — Director of geriatrics
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data (IPD) available to other researchers in a few years.

REFERENCES:
- [Derived] Yang J, Hou L, Wang A, Shang L, Jia X, Xu R, Wang X. Prebiotics improve frailty status in community-dwelling older individuals in a double-blind, randomized, controlled trial. J Clin Invest. 2024 Aug 6;134(18):e176507. doi: 10.1172/JCI176507. PMID 39286985